CLINICAL TRIAL: NCT05078437
Title: Assessment of Medication Optimization in Rural Kentucky Appalachian Patients With Mild Cognitive Impairment or Dementia: The AMOR Kentucky Study
Brief Title: Assessment of Medication Optimization in Rural Kentucky Appalachian Patients With Mild Cognitive Impairment or Dementia
Acronym: AMOR-KY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Daniela Moga (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Northern California Institute of Research and Education (Other)
Responsible Party: Sponsor-Investigator, Daniela Moga, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69305; R24AG064025 (NIH)
Record Dates: First submitted 2021-09-20; First posted 2021-10-14 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Dementia; Mild Cognitive Impairment
Keywords: medication optimization; rural population; dementia; Alzheimer's disease; telemedicine
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Alzheimer Disease | interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment optimization (Experimental): Participants will undergo an evaluation of all the medications taken and changes will be proposed for treatment optimization.
  Interventions: Behavioral: Medication therapy management

INTERVENTIONS:
Behavioral: Medication therapy management — The proposed deprescribing intervention is using a patient-centered framework by: (1) balancing the risks and benefits, and addressing the specific needs of each individual patient, (2) considering the individual patient and the caregiver's preferences and values, and (3) empowering the patient and the caregiver to take responsibility and fully participate in the decision-making process as equal team players.

SUMMARY:
The AMOR-Kentucky study will examine the impact of a pharmacist-physician patient-centered medication therapy management deprescribing intervention to address inappropriate medication use in patients with cognitive impairment in underserved, lower socioeconomic populations in rural Appalachian Kentucky. The results of this study will provide valuable insights on how to expand and implement deprescribing interventions using telemedicine to reduce the prevalence and the associated healthcare costs of medication-related problems in patients with mild cognitive impairment, Alzheimer's disease and other dementias in rural areas throughout the US. The investigators will assess the potential use of telemedicine in this population by performing an initial single arm, unblinded study of the medication therapy management (MTM) describing intervention in rural/underserved Kentucky Appalachian populations with cognitive impairment and/or dementia using potentially inappropriate medications (n=50). Following initial recruitment and clinical evaluation, engaged participants will have their medication list reviewed by a pharmacist-clinician team to identify targets for deprescribing intervention. The intervention will be engaged remotely with the participant and their caregiver, and the MTM team at 4 weeks post initial evaluation, and then reinforced at a 3-month timepoint. This approach will be carried forward through a telemedicine practice at University of Kentucky that is comprised of approximately 500 patient-caregiver dyads throughout rural areas of Appalachian Kentucky.

ELIGIBILITY:
1. 60 years or older,
2. diagnosed with mild cognitive impairment or dementia,
3. using at least one potentially inappropriate medications,
4. living in the community,
5. willing to participate in the study (both the patient and the caregiver)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
This trial will be registered with clinicaltrials.gov and all raw data, stripped of identifiers, will be made available to interested parties and researchers with submission of written request to the study PI not sooner than one year after acceptance and publication of the primary manuscript. There will be no charge for release of the dataset.
Time Frame: not sooner than one year after acceptance and publication of the primary manuscript
Access Criteria: request submitted to the study PI

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Optimization
Started | 16
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Optimization
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 77 [68 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Medication Appropriateness Index
Description: The Medication Appropriateness Index (MAI) is a score based on 10 criteria used to assess the appropriateness of each medication taken by a study participant. Medications are rated as "appropriate", "marginally appropriate", or "inappropriate" based on these ten criteria. Each medication was scored between 0 (appropriate) and the maximum of 18 (inappropriate for all criteria), then the total MAI was obtained by adding the medication specific MAIs for all medications reported by the participant. For each participant, the total MAI is calculated as the sum of the score for all the medications taken by that participant. The minimum is 0 (all medications are appropriate), but there is no maximum because that depends on the number of medications. A decrease in MAI indicates improvement in medication appropriateness.
Time Frame: Baseline and 3 months
Population: For each participant, a change score was calculated based on the MAI at EOS and at baseline. A negative number indicates improvement in appropriateness. The change MAI score is averaged among participants.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Intervention: Participants undergoing the MTM intervention
Arm/Group | Intervention
Number analyzed (Participants) | 12
units on a scale | -5.8 (6.3)

2. Primary Outcome: Participant Satisfaction
Description: Patients will be asked to provide feedback on participation in the deprescribing process.
Time Frame: 6 months
Population: Participants undergoing the MTM intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 13
Participants
  Strongly Agree or Agree | 10
  Neutral | 3

3. Primary Outcome: Connectivity Issues
Description: Participants will be asked to report on any connectivity issues that would impact the appropriate delivery of the intervention using the telemedicine approach. Number of participants that experienced any connectivity issues.
Time Frame: 3 months and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Optimization
Number analyzed (Participants) | 16
Participants | 6

4. Secondary Outcome: Deprescribing Assessments
Description: The revised Patients Attitudes towards deprescribing (rPATD) will assess attitudes towards deprescribing
Time Frame: 6 months
Population: Participants undergoing the MTM intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Optimization
Number analyzed (Participants) | 14
Participants
  Yes or maybe | 11
  No | 3

5. Secondary Outcome: Caregiver Assessment- Zarit
Description: The appraisal of self-care will be used to asses additional outcomes in caregiver. Zarit Burden Interview includes 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden. A score of 17 or more was considered high burden.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Optimization
Number analyzed (Participants) | 15
units on a scale | 1.3 (6.6)

6. Secondary Outcome: Cognitive Function- CDR Global Score
Description: The investigators will use the cognitive battery that is incorporated in the telemedicine assessments to explore the impact of the intervention on cognitive function. Clinical Dementia Rating (CDR) Global Score 0: Normal (unimpaired) cognition; 0.5: MCI due to AD; 1: Mild AD dementia; 2: Moderate AD dementia; 3: Severe AD dementia
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Optimization
Number analyzed (Participants) | 13
score on a scale | 0.2 (0.4)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Information was collected using clinicaltrials.gov definitions during study visit via telehealth
Arm/Group | Treatment Optimization
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Optimization (N=16)
Infection or febrile neutropenia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Optimization (N=16)
allergy/immunology (General disorders) | 2 (2)
gastrointestinal (Gastrointestinal disorders) | 2 (2)
infection or febrile neutropenia (Infections and infestations) | 1 (1)
metabolic/laboratory (Metabolism and nutrition disorders) | 2 (2)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3)
neurology (Nervous system disorders) | 5 (6)
pain (General disorders) | 1 (1)
renal/genitourinary (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT05078437/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT05078437/ICF_000.pdf